CLINICAL TRIAL: NCT06662552
Title: Pulsed Electromagnetic Therapy Versus Whole Body Vibration on Quadriceps Strength Post Burn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Talaat Moustafa Moustafa, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aya-004833
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Pulsed Electromagnetic Field; Whole Body Vibration; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration group (Experimental): Fifteen patients will receive whole body vibration and traditional physical therapy program (splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises) on quadriceps muscle (3 times per week, for 6 weeks), plus medical treatment
  Interventions: Device: whole body vibration using crazy fit machine; Other: traditional physical therapy program
- pulsed electromagnetic field (PEMF) group (Active Comparator): Fifteen patients will receive pulsed electromagnetic field (PEMF) and traditional physical therapy program (splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises) on quadriceps muscle (3 times per week, for 6 weeks), plus medical treatment.
  Interventions: Device: Pulsed electromagnetic field therapy; Other: traditional physical therapy program

INTERVENTIONS:
Device: whole body vibration using crazy fit machine — It will be applied on the whole body All subjects will be asked to stand in a squat position on the vibration platform with the knees bent 90 this position will be chosen because the vertical sinusoidal accelerations of the vibration platform had to be damped by the different muscles around the joints of the lower extremity) ,at a frequency of 30 Hz, 5 - 30 minutes per day, 3 times per week, for 6 weeks, and the physiotherapist will be standing beside the patient
  Arms: whole body vibration group
Device: Pulsed electromagnetic field therapy — EMSCULPT device (BTL Industries Inc., Boston, MA) based on HIFEM technology. It consists of an appliance, motorized bed and solenoids. The appliance will be connected to electrical mains supplying230Vat frequency of 50 or 60 Hz with earth connection, Intensity 0-100. It will be used in the treatment of patient in group "B". Subjects will be positioned in a supine position, and the treatment will be performed by placing the applicator centered over their thigh region (quadriceps muscle's area), for 15 minutes per day, 3 times per week for 6 weeks, the physiotherapist will be sitting beside the patient
  Arms: pulsed electromagnetic field (PEMF) group
Other: traditional physical therapy program — In the form of splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises on quadriceps muscle 15 minutes per day, 3 times per week for 6 weeks.

SUMMARY:
The purpose of the study is to evaluate which is more effective pulsed electromagnetic field therapy or whole-body vibration on quadriceps strength after chronic burn

DETAILED DESCRIPTION:
Severe burn is associated with excessive muscle wasting and atrophy. Muscle wasting is defined as unintentional weight loss of 5%- 10% of muscle mass, and severely burned patients are reported to lose up to 25% of total body mass acutely. (Dirks et al., 2016). These are worsened by deconditioning (eg, prolonged bed rest, immobilization, and inactivity). (Baker et al., 2007).

Furthermore, the need of this study is developed from the lack in the quantitative knowledge and information in the published studies about the effect of pulsed electromagnetic field therapy and whole-body vibration on quadriceps strength after chronic burn.

This study will be designed to provide a guideline about the effect of pulsed electromagnetic field therapy and whole-body vibration on quadriceps strength after chronic burn

ELIGIBILITY:
Inclusion Criteria:

1. Both sex.
2. Their ages will be ranged from 25 to 40 years.
3. Have second degree burn of 10 % to 25 %.
4. Their body mass index (BMI) will not exceed 34.9 Kg/m2.
5. All patients will be clinically and medically stable when attending the study.

Exclusion Criteria:

1. Unstable cardiovascular problems like arrhythmia and heart failure.
2. Diabetes mellitus.
3. Chronic chest disease.
4. Patients on medications affecting muscle power as steroids.
5. Auditory and visual problems.
6. Pregnancy & lactation.
7. Patients with history of epilepsy.
8. Clinically significant peripheral vascular disease.
9. Musculoskeletal or neurological limitation to physical exercise.
10. Any cognitive impairment that interferes with prescribed exercise procedures.
11. Amputation of lower limb.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of change on quadriceps muscle strength using hand-held dynamometer | at baseline and after 6 weeks
  The study involves a bolster positioning to ensure a 35° knee flexion angle, verified using a goniometer. Participants are instructed to maintain their knee in contact with the bolster, with the dominant leg flexed at the hip and knee to stabilize the pelvis. Hips and buttocks are kept flat on the couch, and knee contact is maintained to maintain the angle. Participants are asked to push maximally against the pad to straighten their leg from the knee.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Giza, Egypt